CLINICAL TRIAL: NCT05395442
Title: The Effect of Health Belief Model-Based Web-Based Education on Diabetic Foot Care Knowledge Levels, Behaviors and Self-Efficacy for Individuals With Type 2 Diabetes
Brief Title: Web-based Diabetic Foot Care Training Prepared With the Health Belief Model for Type 2 Diabetes Patients
Acronym: dabe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Yakup SARPDAGI, Research Assistant, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: yakup1
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Diabetic Foot, HBM, Web Based, Self Effectiveness, Self Care
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: A total of 142 people, 71 people in the experimental group and 71 people in the control group, were included in the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, İnvestigator,Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Web-supported diabetic foot care training based on health belief model
  Interventions: Diagnostic Test: Training on web-based diabetic foot care based on the Health Belief Model
- Control Group (No Intervention): No action will be taken.

INTERVENTIONS:
Diagnostic Test: Training on web-based diabetic foot care based on the Health Belief Model — Training on web-based diabetic foot care based on the Health Belief Model will be implemented.Four materials will be used in the research, namely the Introductory Information Form, the Foot Care Behavior Scale, the Diabetic Foot Care Self-Efficacy Scale.
  Arms: Experimental Group

SUMMARY:
Diabetes Mellitus (DM), insulin secretion, insulin action or this It is a chronic metabolic disease characterized by hyperglycemia caused by a defect in both of these factors.

It is an important public health problem that causes organ and function losses due to the complications it creates, negatively affects the life span and quality, and creates a social and economic burden.Diabetic foot, known as an important complication of DM, is an important problem in that it causes deterioration in the quality of life of the patient, frequent and long-term hospitalizations, serious increase in the cost of treatment, lower extremity amputations and increased mortality. As a result of the literature review, it was assumed that the level of knowledge about diabetic foot care could affect diabetic foot care behaviors, self-efficacy and possible diabetic foot complications. In addition to conventional information, a Web-based education based on a health belief model can create awareness in individuals and minimize the risk of diabetic foot ulceration or amputation. The aim of this study is to determine the effect of web-based diabetic foot care training prepared according to SIM on the knowledge levels, self-efficacy and care behaviors of individuals with diabetes.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM), insulin secretion, insulin action or this It is a chronic metabolic disease characterized by hyperglycemia caused by a defect in both of these factors.

It is an important public health problem that causes organ and function losses due to the complications it creates, negatively affects the life span and quality, and creates a social and economic burden.Diabetic foot, known as an important complication of DM, is an important problem in that it causes deterioration in the quality of life of the patient, frequent and long-term hospitalizations, serious increase in the cost of treatment, lower extremity amputations and increased mortality. As a result of the literature review, it was assumed that the level of knowledge about diabetic foot care could affect diabetic foot care behaviors, self-efficacy and possible diabetic foot complications. In addition to conventional information, a Web-based education based on a health belief model can create awareness in individuals and minimize the risk of diabetic foot ulceration or amputation. The aim of this study is to determine the effect of web-based diabetic foot care training prepared according to SIM on the knowledge levels, self-efficacy and care behaviors of individuals with diabetes.

Materials and Methods: This is a randomized controlled experimental study. The research consists of all individuals who are followed up with the diagnosis of type 2 diabetes (1008 people) registered in the Tusba Family Health Center no. Power analysis method was used to determine the sample size of the study. In the power analysis using Cohen's standard effect sizes, it was determined that 128 people, 64 in each group, should be reached in order to reach 80% power at 0.5% effect size, 0.05% margin of error level and 0.95% confidence interval. However, considering that sample loss may occur in the study, 10% more of the calculated sample will be included in the randomization process. In this case, it was determined that a total of 142 people, 71 people in each group, should be reached. In the study, Introductory Information Form, Foot Care Behavior Scale, Diabetic Foot Care Self-Efficacy Scale and Diabetic Foot Information Scale, four materials will be used.The data obtained in this study will be analyzed using the SPSS statistical program (SPSS-22).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 diabetes at least 1 year ago,
* Be between the ages of 18-65,
* Ability to use computer or smartphone,
* With internet access,
* Literate,
* Not having attended training on diabetic foot care,
* Has no disability in answering questions physically, cognitively or spiritually,
* Willingness to participate in research.

Exclusion Criteria:

* Those with a diabetic foot ulcer or amputation,
* Hospitalization in inpatient treatment institutions due to DM or DM complications during the research process,
* Patients with foot deformities (such as overlapping toes),
* Moving to another city during the research process,
* The emergence of any health problem that prevents the person from continuing the research,
* Leaving the research voluntarily.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Pre-Test Data Collection | a month or two
  The pre-test data of the study will be searched by the researcher between June 2022 and July 2022 by obtaining the contact information of the individuals registered in the Van Tusba Family Health Center and included in the study. In the collection of data, the people in the experimental and control groups; Introductory Information Form, Foot Care Behavior Scale, Diabetic Foot Care Self-Efficacy Scale and Diabetic Foot Knowledge Scale" will be applied.
Collection of Post-Test Data | a month or two
  Giving training to the experimental group for 6 weeks with an interval of 2 weeks. The three-month web-based training given by the researcher to the individuals in the experimental group will be completed. After the training is over, a three-month follow-up will be made and post-test data will be collected after 6 months in total. It is planned to collect the final test data in Van Tusba Family Health Center No. 1 between November 2022 and December 2022. In the collection of data, the people in the experimental and control groups; Foot Care Behavior Scale, Diabetic Foot Care Self-Efficacy Scale and Diabetic Foot Knowledge Scale will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Yakup SARPDAĞI, Ph.D, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Van Yüzüncü Yıl Universty, Van, Turkey (Türkiye)